CLINICAL TRIAL: NCT03904901
Title: Influence of Probiotics in Nutritional, Biochemical Profile and Anxiety of Diabetic Cardiopathies With Excessive Weight: a Randomized Clinical Test
Brief Title: Influence of Probiotics in Diabetic Cardiopathies With Excessive Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDallanora
Record Dates: First submitted 2018-10-25; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus Type 2 in Obese; Anxiety; Cardiopathy
MeSH Terms: conditions — Anxiety Disorders; Heart Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics (Active Comparator): Individuals will receive individual capsules containing the daily dose of lyophilized probiotics (Lactobacillus acidophilus, Lactobacillus casei, Lactobacillus lactis, Bifidobacterium lactis and Bifidobacterium bifidum) and will be advised to remain at room temperature, drink with water and drink before bed. Probiotics contain a dose of 10 9 CFU per capsule.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): The placebo product had only the excipient, microcrystalline cellulose, and was identical to the active product in relation to color, shape, size and packaging.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Individuals will receive individual capsules containing the daily dose of lyophilized probiotics (Lactobacillus acidophilus, Lactobacillus casei, Lactobacillus lactis, Bifidobacterium lactis and Bifidobacterium bifidum) and will be advised to remain at room temperature, ingest with water and drink before bed.
  Arms: Probiotics
Dietary Supplement: Placebo — The placebo product had only the excipient, microcrystalline cellulose, and was identical to the active product in relation to color, shape, size and packaging.
  Arms: Placebo

SUMMARY:
Today in Brazil, 6.9% of the population has Diabetes Mellitus 2 (DM2). In the world, there are about 422 million people with DM2. It is a chronic disease of the endocrine system, accounts for 90 to 95% of cases of DM2 and is characterized by defects in insulin action and secretion. Its main cause is linked to obesity and insulin resistance. Obesity is a chronic, multifactorial disease - environmental, nutritional and genetic factors - characterized by excessive accumulation of body fat, and is reaching epidemic proportions, more than 100 million children and 600 million adults worldwide. The number of obese people in Brazil reaches 17.9% of the population.

Rates of obesity and DM2 have increased in the last decades, both diseases being associated with inflammation and specific alterations in the intestinal microbiota. Thus, studies show that the use of probiotics may be associated with reduced body weight and reduced glucose in the bloodstream. Probiotics are living microorganisms that, when administered in suitable dosages, confer benefits to the health of the host. In addition, studies show the relationship of the intestinal microbiota and the emergence of various diseases and demonstrate that probiotics can control inflammatory processes, metabolic dysfunctions, normalization of stress-induced behaviors, regulation of the hypothalamic-pituitary-adrenal axis and neuropsychiatric disorders. Thus, the importance of investigating the ingestion of probiotics in relation to anthropometry, biochemical profile and anxiety in diabetic and overweight individuals with cardiopathy are justified. It is a randomized, double-blind, controlled clinical trial. The study will last 3 months and will occur with 74 adult individuals (between 20 and 60 years) of the SUS outpatient clinic of the Institute of Cardiology of Porto Alegre - RS, of both sexes, with BMI above 25 m² / kg. and less than 40 m² / kg, divided into 2 groups and 37 individuals per group. These patients were: Group A (intervention: n = 37): patient received 1 sachet per day of probiotics Lactobacillus acidophilus, Lactobacillus casei, Lactobacillus lactis, Bifidobacterium lactis and Bifidobacterium bifidum for 90 days and Group B (placebo; n = 37): microcrystalline cellulose, lactose, pregelatinized maize starch. Probiotics will contain a dose of 109 CFU in each strain. The excipients used will be: microcrystalline cellulose.

DETAILED DESCRIPTION:
Probióticos

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years;
* BMI greater than 25 m² / kg and less than 40 m² / kg;
* DM2.

Exclusion Criteria:

* Use of antibiotics or medications for weight loss purposes;
* Use of kefir, yacult;
* Lactose intolerance;
* Inflammatory bowel disease;
* Valvar surgery;
* Use of laxative in the last 3 months;
* Patients participating in other clinical studies.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Control of DM2 | 3 months
  Blood samples were collected fasting (12h overnight) to determine glycemic and hemoglobin (HbA1c)
Anxety | 3 months
  To assess anxiety, was applied by a psychologist to the Beck Scale.
  BAI consists of 21 questions about how the individual has felt in the past week, expressed in common anxiety symptoms (such as sweating and feelings of distress). Each question presents four possible answers, and the one that most closely resembles the individual's mental state must be signaled. The possible answers are:
  Not; Lightly: did not bother me too much; Moderately: it was unpleasant, but I could bear it; Severely: I hardly supported.
  BAI can have a maximum score of 63 and the categories are:
  0-10: minimum degree of anxiety; 11-19: mild anxiety; 20-30 moderate anxiety; Severe anxiety 31-63.

SECONDARY OUTCOMES:
Alteration of serum lipids | 3 months
  Blood samples were collected fasting (fasting of 12h overnight) for glycemia, glycated hemoglobin (HbA1c) in mg / dL, total cholesterol (TC) in mg / dL, high density lipoprotein (HDL-c) in mg / dL, non-HDL in mg / dL and triglycerides in mg / dL. Levels of low-density lipoprotein (LDL in mg / dL) were determined by the Friedewal formula. LDL-c (mg / dL) = TC (mg / dL) - HDL-c (mg / dL) - TG (mg / dL) / 5.
Weight | 3 months
  Body weights were measured using a portable digital scale (Omron brand) without shoes and minimal clothing.
Height | 3 months
  The heights were measured with tape measure fixed to the wall.
BMI | 3 months
  BMI was calculated by dividing body weight (in kilograms) by height (in meters) squared.

CONTACTS AND LOCATIONS:
Overall Officials: Suelen Dallanora, Study Director — Instituto de Cardiologia
Locations (1):
- Suelen Dallanora, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No